CLINICAL TRIAL: NCT03881982
Title: Patient Input Monitoring of Pain in the Emergency Room: Novel Electronic Log (PIMPERNEL). A Randomised Controlled Trial of an Electronic Pain Score Display in Adults in the Emergency Department
Brief Title: A Novel Electronic Method of Collecting Pain Scores in the Emergency Department
Acronym: PIMPERNEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0588; IRAS 210798 (Other: IRAS)
Record Dates: First submitted 2019-01-28; First posted 2019-03-20 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2019-01

CONDITIONS: Pain, Acute
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PIMPERNEL Novel Electronic Log - intervention (Experimental): The display is an electronic version of the 11 point NRS. An audible 'beep' every 15 minutes prompts the patient to record their pain level.
  The display measures 122mm x 30mm x 15mm. Through a wireless connection, the data from the display are transmitted to a display unit (a Nexus tablet).
  Interventions: Other: PIMPERNEL Novel Electronic Log: Pain display can be seen
- PIMPERNEL Novel Electronic Log - control (Other): The display is an electronic version of the 11 point NRS. An audible 'beep' every 15 minutes prompts the patient to record their pain level.
  The display measures 122mm x 30mm x 15mm. Through a wireless connection, the data from the display are transmitted to a display unit (a Nexus tablet).
  Interventions: Other: PIMPERNEL Novel Electronic Log: Pain display is hidden

INTERVENTIONS:
Other: PIMPERNEL Novel Electronic Log: Pain display can be seen — Pain scores are displayed on the screen when the participant presses the corresponding button
  Arms: PIMPERNEL Novel Electronic Log - intervention
Other: PIMPERNEL Novel Electronic Log: Pain display is hidden — Participants press the buttons to record their pain score but the score is not on display (the screen is turned backwards).
  Arms: PIMPERNEL Novel Electronic Log - control

SUMMARY:
Can a novel electronic display of pain be successfully used in the emergency department and does it (1) change analgesic prescription and (2) change amount of pain experienced? Pain is a common symptom in emergency care. As patients are seldom reassessed, staff may not be aware of pain. Currently, members of nursing or medical staff need to ask patients about their pain and record it manually using a visual analogue scale from 0-10.

The new electronic display uses buttons to represent a pain scale from 0 (no pain) to 10 (worst pain). Patients will select the number that best corresponds to their pain every 15 minutes. In the experimental group, the score will be displayed on a screen. In the control group, the score will not be displayed. The investigators will compare the overall amount of pain in both groups, and will look at their pain management (painkillers prescribed). The investigators will also ask patients and staff for their opinions on the display.

The study will include adult patients in the emergency department at Leicester Royal Infirmary with an initial pain score of 5 or more who are able to make a decision about whether to participate. Participants will also need to be likely to stay in the hospital for more than 2 hours to allow the investigators to gather enough useful data. The study will recruit 200 participants. If the study can demonstrate that the monitor is acceptable to patients and staff and results in improved pain management, it is a low cost intervention which could be widely implemented within the NHS. It also has the potential for being used in other areas such as surgical wards. The investigators have previously found that 300-400 patients per week in the department have moderate to severe pain and might therefore benefit from this monitor.

ELIGIBILITY:
Inclusion Criteria:

* adult (18 years and over)
* underlying condition giving rise to significant pain (initial VAS pain score of 5 or more)
* likely to be staying in the hospital for at least 2 hours
* willing and able to give informed consent
* able to understand and speak a good level of English

Exclusion Criteria:

* children (under 18 years)
* patients not willing to undergo routine care (analgesic treatment)
* patients who do not have capacity to consent
* patients who are unwilling or unable to give informed consent
* prisoners
* patients who cannot understand the study information in English
* currently participating in another clinical trial as far as can be determined from information available at the time of assessment
* patients who have a physical or visual disability which will prevent them from holding or using the pain display

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Pain reported by the patient:11 point numerical pain scale | Up to 6 hours
  Data collected from the display using the 11 point numerical pain scale. The area under the curve will be compared between the intervention and control groups. The Numerical Rating Scale is a scale from 0-10 (whole numbers only, where 0 represents 'no pain' and 10 represents 'worst pain ever').

SECONDARY OUTCOMES:
Proportion of possible scores recorded by patients | Up to 6 hours
Comparison of pain recorded on the display (closest minute) with verbal pain assessment at 2 and 4 hours | Up to 6 hours
  The scores recorded by the participants at 2 and 4 hours into their hospital stay will be compared with the scores recorded by nursing staff in the electronic record. The 11 point numerical rating scale is used for both measurements. The Numerical Rating Scale is a scale from 0-10 (whole numbers only, where 0 represents 'no pain' and 10 represents 'worst pain ever').
Understanding the pattern of pain (shape of the curve of pain scores) over the time of the ED stay | Up to 6 hours
Recording time to second dose of analgesia and whether there is a pattern to this | Up to 6 hours
Use of analgesia in intervention and control groups (dose, time prescribed, time administered and name) | Up to 6 hours
  The dose, time prescribed, time administered and name of analgesia given pre-hospital and whilst in hospital will be recorded and a comparison made between the groups. This is a feasibility study only so exact outcome depends upon what data can be collected.
Opinion of patients | Up to 6 hours
  Uses a short (4 question) questionnaire designed for this study. Questions on ease of use, whether the monitor is a good idea, whether participants would use it again in the future and whether it improved their experience as a patient, plus a comments box.
  Questions: 1) How easy was it to use the pain monitor? (very easy, easy, no opinion, difficult, very difficult) 2) I think that the pain monitor is a good idea (strongly agree, agree, no opinion, disagree, strongly disagree) 3) I would use the monitor again in the future (strongly agree, agree, no opinion, disagree, strongly disagree) 4) The pain monitor improved my experience as a patient (strongly agree, agree, no opinion, disagree, strongly disagree)
Opinion of staff (including their opinion of whether patients press the button for reasons other than pain) | Up to 6 hours
  Short (4 question) questionnaire designed for the study. Questions on whether the display is practical to use in the Emergency Department, whether they think it is a good idea, whether it is likely to improve the patient experience and whether a patient used the display to get their attention for a reason other than pain. Also has a comments box.
  Questions: 1) The pain display is practical to use in the Emergency Department (strongly agree, agree, no opinion, disagree, strongly disagree) 2) I think that the pain display is a good idea (strongly agree, agree, no opinion, disagree, strongly disagree) 3) The pain display is likely to improve the patient experience (strongly agree, agree, no opinion, disagree, strongly disagree) 4) A patient used the pain display to get my attention for a reason other than pain (yes, not sure, no)
Opinion of researchers regarding any likely stratification needs | Up to 6 hours
  Subjective opinion of researchers having completed the study on whether stratification would be required in future studies. No specific measurement used.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J Coats, Prof, Principal Investigator — University of Leicester
Locations (1):
- Leicester Royal Infirmary, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
We are collecting feasibility data only in this trial.

REFERENCES:
- [Background] Johnston CC, Gagnon AJ, Fullerton L, Common C, Ladores M, Forlini S. One-week survey of pain intensity on admission to and discharge from the emergency department: a pilot study. J Emerg Med. 1998 May-Jun;16(3):377-82. doi: 10.1016/s0736-4679(98)00012-2. PMID 9610963
- [Background] Cordell WH, Keene KK, Giles BK, Jones JB, Jones JH, Brizendine EJ. The high prevalence of pain in emergency medical care. Am J Emerg Med. 2002 May;20(3):165-9. doi: 10.1053/ajem.2002.32643. PMID 11992334
- [Background] Ducharme J, Barber C. A prospective blinded study on emergency pain assessment and therapy. J Emerg Med. 1995 Jul-Aug;13(4):571-5. doi: 10.1016/0736-4679(95)80023-9. PMID 7594383
- [Background] Todd KH, Ducharme J, Choiniere M, Crandall CS, Fosnocht DE, Homel P, Tanabe P; PEMI Study Group. Pain in the emergency department: results of the pain and emergency medicine initiative (PEMI) multicenter study. J Pain. 2007 Jun;8(6):460-6. doi: 10.1016/j.jpain.2006.12.005. Epub 2007 Feb 15. PMID 17306626
- [Background] Motov SM, Khan AN. Problems and barriers of pain management in the emergency department: Are we ever going to get better? J Pain Res. 2008 Dec 9;2:5-11. PMID 21197290
- [Background] Rupp T, Delaney KA. Inadequate analgesia in emergency medicine. Ann Emerg Med. 2004 Apr;43(4):494-503. doi: 10.1016/j.annemergmed.2003.11.019. PMID 15039693
- [Background] Loryman B, Davies F, Chavada G, Coats T. Consigning "brutacaine" to history: a survey of pharmacological techniques to facilitate painful procedures in children in emergency departments in the UK. Emerg Med J. 2006 Nov;23(11):838-40. doi: 10.1136/emj.2006.034140. PMID 17057133
- [Background] Brown JC, Klein EJ, Lewis CW, Johnston BD, Cummings P. Emergency department analgesia for fracture pain. Ann Emerg Med. 2003 Aug;42(2):197-205. doi: 10.1067/mem.2003.275. PMID 12883507
- [Background] Stahmer SA, Shofer FS, Marino A, Shepherd S, Abbuhl S. Do quantitative changes in pain intensity correlate with pain relief and satisfaction? Acad Emerg Med. 1998 Sep;5(9):851-7. doi: 10.1111/j.1553-2712.1998.tb02811.x. PMID 9754496
- [Background] FitzGerald G, Jelinek GA, Scott D, Gerdtz MF. Emergency department triage revisited. Emerg Med J. 2010 Feb;27(2):86-92. doi: 10.1136/emj.2009.077081. PMID 20156855
- [Background] Telfer P, Criddle J, Sandell J, Davies F, Morrison I, Challands J. Intranasal diamorphine for acute sickle cell pain. Arch Dis Child. 2009 Dec;94(12):979-80. doi: 10.1136/adc.2008.138875. Epub 2009 Mar 25. PMID 19321506
- [Background] France J, Smith S, Smith L. The College of Emergency Medicine Best Practice Guideline: Management of Pain in Adults. 2014.
- [Background] Menendez ME, Bot AG, Hageman MG, Neuhaus V, Mudgal CS, Ring D. Computerized adaptive testing of psychological factors: relation to upper-extremity disability. J Bone Joint Surg Am. 2013 Oct 16;95(20):e149. doi: 10.2106/JBJS.L.01614. PMID 24132364
- [Background] Smith JE, Rockett M, Squire R, Hayward CJ, Creanor S, Ewings P, Barton A, Pritchard C, Benger JR. PAin SoluTions In the Emergency Setting (PASTIES); a protocol for two open-label randomised trials of patient-controlled analgesia (PCA) versus routine care in the emergency department. BMJ Open. 2013 Feb 14;3(2):e002577. doi: 10.1136/bmjopen-2013-002577. Print 2013. PMID 23418302